CLINICAL TRIAL: NCT06340997
Title: Impact of Percutaneous Transvenous Mitral Commissurotomy on The Left Atrial Appendage Function in Patients With Mitral Stenosis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ali Ismail, Resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Mitral Stenosis
Record Dates: First submitted 2023-12-14; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Mitral Stenosis
MeSH Terms: conditions — Mitral Valve Stenosis | interventions — Echocardiography, Transesophageal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with mitral stenosis (Other)
  Interventions: Device: Transesophageal echocardiography

INTERVENTIONS:
Device: Transesophageal echocardiography — * D.Echocardiography(Transthoracic and transesophageal):
  * 2D echocardiography (to detect LA function, severity of MS and Wilkins score).
  The following conventional parameters were measured :
  * left atrial volume index (LAVi), and left ventricular ejection fraction (LVEF) by modified biplane Simpson's rule , left atrial emptying fraction calculated as (LAVi max-LAVi min)/LAVi max × 100 ,]degree of concomitant mitral regurgitation. The maximum and minimum LAA areas were measured by planimetry. LAA area change (%) was calculated using the following formula: LAA area change = [(maximal LAA area-minimal LAA area)/maximal LAA area] × 100.
  * Transesophageal echocardiogram (TEE) (to detect LAA function) .
  * LAA flow velocity patterns by pulsed-wave Doppler
  * Early diastolic emptying velocity
  * Late diastolic emptying velocity or LAA contraction flow
  * LAA filling velocity
  * Systolic reflection waves
  * Two-Dimensional- LAA fractional area change (LAAAC%)

SUMMARY:
• Evaluation of the effect of PTMC on LAA function by TEE at least one month after the procedure and its effectiveness in prevention of thrombi formation and cerebrovascular complications.

DETAILED DESCRIPTION:
* Mitral stenosis (MS) is a disabling disease that limits the normal physical abilities of patients and considered as a major reason for hospital admissions . The leading cause of MS globally is rheumatic heart disease(RHD), which remains common in economically developing countries and continues to be a significant cause of morbidity and mortality.
* Chronic pressure and volume overload imposed by MS causes left atrial (LA) and Left Atrial Appendage (LAA) dysfunction leading to reduced blood flow velocities thereby producing stasis of blood, reduced LA and LAA ejection fraction and atrial fibrillation (AF).
* These factors predispose to formation of LA and LAA thrombi in MS and result in thromboembolic episodes. Risk of cerebrovascular accident (CVA) is increased approximately five-fold in non-rheumatic AF and 17-fold in patients with MS with AF. Even patients of MS in sinus rhythm with depressed LA and LAA function are at increased risk of CVA. Assessment of LAA function is helpful in predicting the risk of thromboembolism .
* PTMC can improve the function of the LAA by reducing the left atrial pressure and increasing the blood flow through the mitral valve.
* Echocardiography, particularly transesophageal echocardiography (TEE), is currently the modality of choice for evaluation of the LAA. Transesophageal echocardiography (TEE) allows semi-invasive, highly accurate imaging of the functional efficiency of LAA by LAA Doppler and Doppler tissue imaging (DTI) .
* MS causes decreased LAA Doppler and DTI velocities in patients even with sinus rhythm . So, this study aims to evaluate effect of successful PTMC on LAA function by TEE Doppler and DTI (doppler tissue imaging).
* Fractional area change (FAC): The FAC is a measure of the percentage of change in the area of the LAA during systole. A higher FAC indicates a more contractile LAA.

ELIGIBILITY:
Inclusion Criteria:

* • Patient eligible for PTMC as anatomical characteristics àpatient with sever MS (area 1.5cm2, echocardiographic score (Wilkins score ≤ 8, Cormier score 1 and 2 …), contraindication or high risk to surgical MVR.

Exclusion Criteria:

* Patient with mitral regurgitation more than grade II .
* Patient not eligible to PTMC.
* Patient with severe heart failure (NHYA class IV) .
* Patient with previous Cerebrovascular accident .
* Patient with contraindication to TEE ( esophageal disease like stricture , diverticuli, varices, …, uncooperative patient )

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Impact of Percutaneous Transvenous Mitral Commissurotomy on The Left Atrial Appendage Function in Patients with Mitral Stenosis. | basline
  Assessment of left atrial appendage function pre and post PTMC. This assessment will be carried out through echocardiography by describing if it contains thrombus or not.

SECONDARY OUTCOMES:
Prevention of left atrial appendage thrombus. | basline
  Improvement of LAA function and its clinical repercussion in preventing thrombus formation and consequently cerebrovascular accidents by follow up LAA function and whether thrombus is formed or not.